CLINICAL TRIAL: NCT03515408
Title: Individualized Precise Localization of rTMS on Precentral and Parietal Gyrus and Its Effects on Dorsal Anterior Cingulate Cortex
Brief Title: Individualized Precise Localization of rTMS on Precentral and Parietal Gyrus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Yu-Feng ZANG, Professor, Hangzhou Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HZNU_sustainded_attention_rTMS
Record Dates: First submitted 2018-04-06; First posted 2018-05-03 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: fMRI; rTMS; functional connectivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Real rTMS (motor area) (Experimental): Real rTMS targeting motor area for 30 min
  Interventions: Device: rTMS
- Real rTMS (parietal gyrus) (Experimental): Real rTMS targeting parietal gyrus for 30 min
  Interventions: Device: rTMS
- Real rTMS (both brain area) (Experimental): Real rTMS targeting motor area and parietal gyrus for 15 min, separately
  Interventions: Device: rTMS
- Sham rTMS (Sham Comparator): Sham rTMS targeting motor area and parietal gyrus for 15 min, separately
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — The 10-Hz stimulation is delivered at 100% of the subject's resting motor threshold via 60 trains of 3-s 10-Hz rTMS (30 pulses with 27-s duration per train).

SUMMARY:
Attention deficit hyperactivity disorder (ADHD) patients have some problem with sustained attention. The dorsal anterior cingulate cortex (dACC) plays a key role for attention control. It has been found that the dACC has strong functional connectivity with ipsilateral motor area and parietal gyrus. Repetitive Transcranial Magnetic Stimulation (rTMS) is a sage and painless technique to activate cortical areas. The deep brain structure can be activated via stimulating superficial cortex by rTMS. For investigating the mechanism of sustained attention, this project is using functional magnetic resonance imaging (fMRI) to individualize the precise localization in motor area and parietal gyrus, and combining rTMS to activate the dACC.

DETAILED DESCRIPTION:
Healthy subject is recruiting in this project. High rTMS will be performed. The 10-Hz stimulation is delivered at 100% of the subject's resting motor threshold via 60 trains of 3-s 10-Hz rTMS (30 pulses with 27-s duration per train).

ELIGIBILITY:
Inclusion Criteria:

* There are activation in dACC, motor area and parietal gyrus during the task fMRI
* The head motion less than 2 mm in translation or 2 degrees in rotation in any direction during the resting-state fMRI

Exclusion Criteria:

* Without any neuropsychiatric conditions
* No head injury or history of epilepsy
* Not on any medications

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-04-08 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
degree of enhanced neuro-activity associated with target-specific treatment | through study completion, an average of 1 year
  amplitude of low frequency fluctuation

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Feng Zang, M.D., Principal Investigator — Hangzhou Normal University
Locations (1):
- Hangzhou Normal University,Center for Cognition and Brain Disorder, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The IPD data cannot be shared with other researchers right now. We will shared it two years later.

REFERENCES:
- [Result] Eldaief MC, Halko MA, Buckner RL, Pascual-Leone A. Transcranial magnetic stimulation modulates the brain's intrinsic activity in a frequency-dependent manner. Proc Natl Acad Sci U S A. 2011 Dec 27;108(52):21229-34. doi: 10.1073/pnas.1113103109. Epub 2011 Dec 12. PMID 22160708
- [Result] Wang JX, Rogers LM, Gross EZ, Ryals AJ, Dokucu ME, Brandstatt KL, Hermiller MS, Voss JL. Targeted enhancement of cortical-hippocampal brain networks and associative memory. Science. 2014 Aug 29;345(6200):1054-7. doi: 10.1126/science.1252900. PMID 25170153
- [Result] Wang J, Yang N, Liao W, Zhang H, Yan CG, Zang YF, Zuo XN. Dorsal anterior cingulate cortex in typically developing children: Laterality analysis. Dev Cogn Neurosci. 2015 Oct;15:117-29. doi: 10.1016/j.dcn.2015.10.002. PMID 26602957